CLINICAL TRIAL: NCT03154307
Title: Repeated TMS at Low Frequencies to Reduce Seizure Occurrence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Recruitment
Sponsor: Baptist Health South Florida (Other)
Collaborators: U.S. National Science Foundation (U.S. Federal Agency); Florida International University (Other)
Responsible Party: Principal Investigator, Alberto Pinzon, M.D., Neurologist, Medical Director, Baptist Health Epilepsy Program, Baptist Health South Florida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-135
Record Dates: First submitted 2017-05-10; First posted 2017-05-16 (Actual); Results first posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-05

CONDITIONS: Epilepsy; Status Epilepticus; Epilepsia Partialis Continua; Epilepsia Partialis Continua, Refractory (Medically)
MeSH Terms: conditions — Epilepsy; Status Epilepticus; Epilepsia Partialis Continua

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and outcomes assessor will be masked in the 3 arms of the long-term protocol. However, the short-term arm will be open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Group 1: Weekly TMS (Experimental): LF-rTMS intervention for 2 weeks (5 days per week for total of 10 days) , LF-rTMS 1 session/week for 1 month (4 days), and LF-rTMS 1 session/month for 11 months
  Interventions: Device: Low frequency repeated TMS (LF-rTMS)
- Group 2: Monthly TMS (Experimental): LF-rTMS intervention for 2 weeks (5 days per week for total of 10 days), LF-rTMS 1 session/month for 12 months
  Interventions: Device: Low frequency repeated TMS (LF-rTMS)
- Group 3: Sham TMS (Sham Comparator): Sham LF-rTMS for 2 weeks (5 days per week for a total of 10 days), sham LF-rTMS 1 session/week for 1 month (4 days), and sham LF-rTMS 1 session/month for 1 month. After the sham stimulation real LF-rTMS intervention sessions will be delivered as follows: 50% of placebo group will follow group 1 protocol and the other 50% will follow group 2 protocol
  Interventions: Device: Low frequency repeated TMS (LF-rTMS)
- Short-term protocol (Experimental): LF-rTMS intervention daily for up to 5 days in medically refractory status epilepticus participants only
  Interventions: Device: Low frequency repeated TMS (LF-rTMS)

INTERVENTIONS:
Device: Low frequency repeated TMS (LF-rTMS) — Each patient will then begin treatment with 14 minute sessions of 1 Hz rTMS or sham rTMS, 120% minimum threshold (MT), and 800 stimuli on the position of the calculated 3D source using EEG, MRI, and digitized electrode locations. Two different timelines of delivering the rTMS will be compared against a sham/delayed treatment group.

SUMMARY:
Perform non-invasive neuro-navigated repeated Transcranial Magnetic Stimulation (rTMS) at low frequencies (LF) with the intent to reduce the occurrence of seizures over time (long-term protocol). Seizure reduction and improvements in the quality of life in patients with epilepsy will be associated with increased cortical inhibition resulting from the LF-rTMS sessions over time. This procedure using rTMS at low frequencies (LF-rTMS) between 0.5 and 1 Hz is a safe and painless method for noninvasive focal cortical brain stimulation, which will be evaluated in its efficacy at reducing/suppressing seizures. Accordingly, we propose a clinical trial in patients with epilepsy to test whether LF-rTMS can improve seizure suppression. The location of the presumed 3D source in the brain will be stimulated for few minutes (10 to 15 min.). With the same rTMS modality, we will also perform motor threshold mapping in conjunction with its fully integrated and compatible electroencephalography (EEG) module. Up to 100 individuals 18 to 80 years with epilepsy will be enrolled.

In addition, a short-term protocol has been added to test whether LF-rTMS can reduce or suppress status epilepticus in medically refractory participants.

DETAILED DESCRIPTION:
Long term protocol: Perform non-invasive neuro-navigated repeated Transcranial Magnetic Stimulation (rTMS) at low frequencies (LF) with to reduce the occurrence of seizures over time. Seizure reduction and improvements in the quality of life in patients with epilepsy will be associated with increased cortical inhibition resulting from the LF-rTMS sessions over time. This procedure using rTMS at low frequencies (LF-rTMS) between 0.5 and 1 Hz is a safe and painless method for noninvasive focal cortical brain stimulation, which will be evaluated in its efficacy at reducing/suppressing seizures. Accordingly, we propose a clinical trial in patients with epilepsy to test whether LF-rTMS can improve seizure suppression. The location of the presumed 3D source in the brain will be stimulated for few minutes (10 to 15 min.). Using a double-blinded, sham-controlled design, we will enroll up to 100 participants aged 18-80 with focal and generalized retractable epilepsy. Baseline data will include a detailed seizure diary over 4 weeks, psychometric testing/neuropsychology evaluation, and 20-minute EEG recordings. Each patient will then begin treatment with 14 minute sessions of 1 Hz rTMS or sham rTMS, 120%MT, and 800 stimuli on the position of the calculated 3D source using EEG, MRI, and digitized electrode locations. The protocol will be divided in 3 groups (Groups 1, 2 and 3) as follows:

* Groups 1, 2, and 3: LF-rTMS for 2 weeks (5 days per week for total of 10 days).
* Group 1: protocol total duration: 1 year: LF-rTMS 1 session/week for 1 month (4 days), and LF-rTMS 1 session/month for 11 months
* Group 2: protocol total duration: 1 year: LF-rTMS 1 session/month for 12 months
* Group 3 (placebo protocol, total duration: 1 year): LF-rTMS 1 session/week for 1 month (4 days); and LF-rTMS 1session/month.

During each session EEG may be recorded. Also, we will obtain the number, frequency, and duration of seizure events from an ongoing seizure diary. Psychometric testing will be performed at the beginning of study, 3 months, and at the end of the study. Thus, each patient will have rTMS testing, psychometrics, and EEG recordings. With the same rTMS modality, we will also perform motor threshold mapping in conjunction with its fully integrated and compatible electroencephalography (EEG) module.

Short-term protocol: Use LF-rTMS protocol as described but for up to 5 days in 10 participants with medically refractory status epilepticus. During each session EEG will be recorded.

ELIGIBILITY:
Long-term protocol:

Inclusion Criteria:

* Experience ≥ 3 seizures/month in the month prior to starting study (any type of seizure will count)
* No status epilepticus in the last 12 months
* No change in medication in last 30 days

Exclusion Criteria:

* Presence of implanted electronic devices (e.g., pacemaker, medication pump, brain or vagus nerve stimulator, cochlear implant)
* Presence of intracranial metal (e.g., aneurysm clip)
* Unable to cooperate with non-sedated, navigated TMS testing

Short-term protocol:

Inclusion Criteria:

* Epilepsia partialis continua or status epilepticus
* At least 2 medications failed
* At least 24 hours of acute phase

Exclusion Criteria:

* Presence of implanted electronic devices (e.g., pacemaker, medication pump, brain or vagus nerve stimulator, cochlear implant)
* Presence of intracranial metal (e.g., aneurysm clip)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Pinzon, M.D., Ph.D., Principal Investigator — Baptist Health South Florida
Locations (1):
- Baptist Hospital of Miami, Miami, Florida, United States

REFERENCES:
- [Background] Kobayashi M, Pascual-Leone A. Transcranial magnetic stimulation in neurology. Lancet Neurol. 2003 Mar;2(3):145-56. doi: 10.1016/s1474-4422(03)00321-1. PMID 12849236
- [Background] Hallett M. Transcranial magnetic stimulation and the human brain. Nature. 2000 Jul 13;406(6792):147-50. doi: 10.1038/35018000. PMID 10910346
- [Background] Rossini PM, Rossi S. Transcranial magnetic stimulation: diagnostic, therapeutic, and research potential. Neurology. 2007 Feb 13;68(7):484-8. doi: 10.1212/01.wnl.0000250268.13789.b2. PMID 17296913
- [Background] Siebner HR, Hartwigsen G, Kassuba T, Rothwell JC. How does transcranial magnetic stimulation modify neuronal activity in the brain? Implications for studies of cognition. Cortex. 2009 Oct;45(9):1035-42. doi: 10.1016/j.cortex.2009.02.007. Epub 2009 Mar 3. PMID 19371866
- [Background] Udupa K, Sathyaprabha TN, Thirthalli J, Kishore KR, Raju TR, Gangadhar BN. Modulation of cardiac autonomic functions in patients with major depression treated with repetitive transcranial magnetic stimulation. J Affect Disord. 2007 Dec;104(1-3):231-6. doi: 10.1016/j.jad.2007.04.002. Epub 2007 May 8. PMID 17490754
- [Background] Fox MD, Liu H, Pascual-Leone A. Identification of reproducible individualized targets for treatment of depression with TMS based on intrinsic connectivity. Neuroimage. 2013 Feb 1;66:151-60. doi: 10.1016/j.neuroimage.2012.10.082. Epub 2012 Nov 7. PMID 23142067
- [Background] Plewnia C, Pasqualetti P, Grosse S, Schlipf S, Wasserka B, Zwissler B, Fallgatter A. Treatment of major depression with bilateral theta burst stimulation: a randomized controlled pilot trial. J Affect Disord. 2014 Mar;156:219-23. doi: 10.1016/j.jad.2013.12.025. Epub 2013 Dec 28. PMID 24411682

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: Weekly TMS | Group 2: Monthly TMS | Group 3: Sham TMS | Short-term Protocol
Started | 2 | 0 | 0 | 0
Completed | 1 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated due to low enrollment. No analysis was completed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Weekly TMS | Group 2: Monthly TMS | Group 3: Sham TMS | Short-term Protocol | Total
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 0 | 0 | 1
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 1 | 0 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 1 | 0 | 0 | 0 | 1
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Baseline Seizure frequency per week [Mean (Full Range); unit: seizures per week] — Data was collected by caregiver for 2-weeks prior to receiving rTMS treatment to establish a weekly seizure frequency. Population: Baseline data was not fully collected for 1 patient who withdrew from the study.
  seizures per week | 37 [31 to 43] |  |  |  | 37 [31 to 43]
Scalp EEG Functional Connectivity for Alpha Hz [Number; unit: Standardized EEG connections] — Baseline Standardized functional scalp EEG connection per of region (anterior, posterior, right, left). Calculations required EEG electrode activity of 80% for a minimum of 20 epochs to be included. All area electrode counts were then divided by the threshold providing a normalized value per brain region.
  Standardized EEG connections
    Anterior | 2.44 |  |  |  | 2.44
    Posterior | 1.0 |  |  |  | 1.0
    Right | 2.425 |  |  |  | 2.425
    Left | 0.63 |  |  |  | 0.63
Baseline Seizure Duration Proxy for Seizure Severity [Mean (Standard Deviation); unit: seconds] — Care provider journaled the seizure duration over the course of a 2-week period prior to receiving rTMS treatment to establish baseline seizure severity.
  seconds | 26.08 (28.97) |  |  |  | 26.08 (28.97)
Abductor Pollicis Brevis (APB)-evoked response threshold [Number; unit: percentage of max Telsa] — The motor evoked potential (MEP) will be calculated using the Nexstim system's 6-channel EMG module (SR=1450 Hz, cut-off frequency of 350 Hz for the low pass filter) as the APB is stimulated to find the threshold for each individual. Listed values represent the percentage of the maximum Tesla output of the Nexstim system.
  percentage of max Telsa | 40 |  |  |  | 40
Interhemispheric EEG Asymmetry Ratio for Alpha power [Number; unit: Ratio] — Expresses the ratio of laterality for the corresponding electrode pairs between the left and right hemispheres, where the left hemisphere electrodes are divided by the right hemisphere electrodes.
  Ratio | 1.26 |  |  |  | 1.26
Intrahemispheric EEG Asymmetry Ratio for Alpha power [Number; unit: Ratio] — Expresses the asymmetry power ratio for the corresponding electrode pairs between the posterior and anterior brain regions, where the left posterior electrodes are divided by the anterior electrodes.
  Ratio | 1.28 |  |  |  | 1.28

OUTCOME MEASURES:

1. Primary Outcome: Average Weekly Seizure Frequency
Description: Seizure frequency was recorded by the caregiver in a journal at weeks 6 and 7 post rTMS treatment.
Time Frame: 6 and 7 weeks post rTMS treatment
Population: Post rTMS seizure journal
Measure: Mean (Full Range); unit: average seizure frequency per week
Units Other Than Participants: seizures
Arm/Group | Group 1: Weekly TMS | Group 2: Monthly TMS | Group 3: Sham TMS | Short-term Protocol
Number analyzed (Participants) | 1 | 0 | 0 | 0
Number analyzed (seizures) | 44 | 0 | 0 | 0
average seizure frequency per week | 22 [21 to 23] |  |  |

2. Primary Outcome: Scalp EEG: Number of Interictal Epileptiform Discharges
Description: Interictal discharges are common in those with epilepsy and tends to decrease with treatment.
Time Frame: From start of intervention through 5 days of treatment
Population: No interictal discharges were observed during baseline or post-treatment.
Measure: Number; unit: Interictal discharges
Arm/Group | Group 1: Weekly TMS | Group 2: Monthly TMS | Group 3: Sham TMS | Short-term Protocol
Number analyzed (Participants) | 1 | 0 | 0 | 0
Interictal discharges | 0 |  |  |

3. Primary Outcome: Seizure Duration Proxy for Seizure Severity
Description: Care provider journaled the seizure duration over the coure of a 2-week period beginning on week 6 post rTMS treatment.
Time Frame: 6-7-weeks post rTMS treatment
Population: Post rTMS seizure journal
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: seizures
Arm/Group | Group 1: Weekly TMS | Group 2: Monthly TMS | Group 3: Sham TMS | Short-term Protocol
Number analyzed (Participants) | 1 | 0 | 0 | 0
Number analyzed (seizures) | 44 | 0 | 0 | 0
seconds | 34.54 (26.14) |  |  |

4. Secondary Outcome: Interhemispheric EEG Asymmetry Ratio for Alpha Power
Description: Expresses the ratio of laterality for the corresponding electrode pairs between the left and right hemispheres, where the left hemisphere electrodes are divided by the right hemisphere electrodes.
Time Frame: 8-weeks Post rTMS Treatment
Population: left hemisphere electrodes are divided by the right hemisphere electrodes
Measure: Number; unit: Ratio
Arm/Group | Group 1: Weekly TMS | Group 2: Monthly TMS | Group 3: Sham TMS | Short-term Protocol
Number analyzed (Participants) | 1 | 0 | 0 | 0
Ratio | 0.45 |  |  |

5. Secondary Outcome: Scalp EEG Functional Connectivity for Alpha Hz
Description: Standardized functional scalp EEG connection per of region (anterior, posterior, right, and left). Calculations required EEG electrode activity of 80% for a minimum of 20 epochs to be included. All area electrode counts were then divided by the threshold providing a normalized value per brain region. Scalp EEG connectivity was collected 8-weeks post rTMS treatment.
Time Frame: 8-weeks Post rTMS Treatment
Population: Data was based on standardized threshold of 80% across 20 Epochs
Measure: Number; unit: Standardized EEG connections
Arm/Group | Group 1: Weekly TMS | Group 2: Monthly TMS | Group 3: Sham TMS | Short-term Protocol
Number analyzed (Participants) | 1 | 0 | 0 | 0
Standardized EEG connections
  Anterior | 0.4 |  |  |
  Posterior | 0.455 |  |  |
  Right | 0.375 |  |  |
  Left | 0.255 |  |  |

6. Secondary Outcome: Abductor Pollicis Brevis (APB)-Evoked Response Threshold
Description: The motor evoked potential (MEP) will be calculated using the Nexstim system's 6-channel EMG module (SR=1450 Hz, cut-off frequency of 350 Hz for the low pass filter) as the APB is stimulated to find the threshold for each individual. Listed values represent the percentage of the maximum Tesla output of the Nexstim system.
Time Frame: 8-weeks Post rTMS treatment
Population: Post APB-evoked response was not collected, therefore cannot be analyzed.
Arm/Group | Group 1: Weekly TMS | Group 2: Monthly TMS | Group 3: Sham TMS | Short-term Protocol
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Treatment Response Rate
Description: Count of subjects whose seizure frequency decreased by 50% after rTMS treatment
Time Frame: 8-weeks post rTMS treatment
Population: The only subject to complete the study was assigned the group 1. Due to lack of enrollment no subjects were assigned to group 2, 3, or the short-term group.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Weekly TMS | Group 2: Monthly TMS | Group 3: Sham TMS | Short-term Protocol
Number analyzed (Participants) | 1 | 0 | 0 | 0
Participants
  Responder (> 50%) | 0 |  |  |
  Non-Responder (<50%) | 1 |  |  |

8. Secondary Outcome: Intrahemispheric EEG Asymmetry Ratio for Alpha Power
Description: Expresses the asymmetry power ratio for the corresponding electrode pairs between the posterior and anterior brain regions, where the left posterior electrodes are divided by the anterior electrodes.
Time Frame: 8-weeks Post rTMS Treatment
Population: left posterior electrodes are divided by the anterior electrodes
Measure: Number; unit: Ratio
Arm/Group | Group 1: Weekly TMS | Group 2: Monthly TMS | Group 3: Sham TMS | Short-term Protocol
Number analyzed (Participants) | 1 | 0 | 0 | 0
Ratio | 0.095 |  |  |

ADVERSE EVENTS:
Time Frame: 1 year
Description: Study was terminated due to low enrollment.
Arm/Group | Group 1: Weekly TMS | Group 2: Monthly TMS | Group 3: Sham TMS | Short-term Protocol
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/07/NCT03154307/Prot_SAP_000.pdf